CLINICAL TRIAL: NCT00259012
Title: A Multicenter, Randomized, Open Label, Single and Multiple Dose Study of the Pharmacokinetics and Pharmacodynamics of 2 Dose Levels of Pantoprazole Sodium Enteric-Coated Spheroid Suspension in Infants Aged 1 Through 11 Months With Presumed GERD
Brief Title: Study Evaluating Pantoprazole Sodium Enteric-Coated Spheroid Suspension In Infants With Presumed GERD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Nycomed (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3001B3-333, 3001B3-335
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Results first posted 2010-05-07 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD; Infant
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose (Active Comparator)
  Interventions: Drug: pantoprazole sodium enteric-coated spheroid suspension
- High dose (Active Comparator)
  Interventions: Drug: pantoprazole sodium enteric-coated spheroid suspension

INTERVENTIONS:
Drug: pantoprazole sodium enteric-coated spheroid suspension — pediatric suspension taken daily x 7 days

SUMMARY:
The purpose of this study is to characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profiles to determine the safety and tolerability of single and multiple doses of pantoprazole in infants aged 1 through 11 months.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 44 weeks beyond neonatal period but less than 12 months
* Presumptive diagnosis of GERD
* Weight greater than 2.5 kg but less than 15 kg

Exclusion Criteria:

* History of gastrointestinal (GI) disorders, ie, unrepaired tracheal esophageal fistula, GI malabsorption
* Clinically significant medical or surgical abnormalities

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2005-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Switzerland, med@wyeth.com
Locations (31):
- United States (16):
  - Little Rock, Arkansas
  - Loma Linda, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Pensacola, Florida
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Jackson, Mississippi
  - Kansas City, Missouri
  - New York, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Temple, Texas
- Brisbane, Australia
- Belgium (3):
  - Antwerp
  - Brussels
  - Ghent
- Paris, France
- Germany (2):
  - Aachen
  - Osnabrück
- Italy (3):
  - Brescia
  - Naples
  - Roma
- Poland (4):
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
- Zurich, Switzerland

REFERENCES:
- [Derived] Tammara BK, Sullivan JE, Adcock KG, Kierkus J, Giblin J, Rath N, Meng X, Maguire MK, Comer GM, Ward RM. Randomized, open-label, multicentre pharmacokinetic studies of two dose levels of pantoprazole granules in infants and children aged 1 month through <6 years with gastro-oesophageal reflux disease. Clin Pharmacokinet. 2011 Aug;50(8):541-50. doi: 10.2165/11591900-000000000-00000. PMID 21740077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited February 2006 to January 2008.
Pre-assignment Details: Patients were screened for seven days.
Groups:
- Low Dose Pantoprazole (0.6 mg/kg): Patients weighing 2.5 to <7 kg received pantoprazole sodium enteric-coated spheroid suspension daily 2.5 mg. Patients weighing ≥7 to ≤15 kg received pantoprazole sodium enteric-coated spheroid suspension daily 5 mg. This dosing corresponds to approximately 0.6 mg/kg.
- High Dose Pantoprazole (1.2 mg/kg): Patients weighing 2.5 to <7 kg received pantoprazole sodium enteric-coated spheroid suspension daily 5 mg. Patients weighing ≥7 to ≤15 kg received pantoprazole sodium enteric-coated spheroid suspension daily 10 mg. This dosing corresponds to approximately 1.2 mg/kg.
Period: Overall Study
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Started | 33 | 34
Completed | 31 | 30
Not Completed | 2 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg) | Total
Number analyzed (Participants) | 33 | 34 | 67
Age Continuous [Mean (Standard Deviation); unit: months] | 5.98 (2.98) | 5.91 (3.42) | 5.94 (3.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28.0
  Male | 20 | 19 | 39.0

OUTCOME MEASURES:

1. Primary Outcome: Peak Concentration (Cmax)
Description: Pharmacokinetic (PK) parameters, including peak plasma concentration, were determined following a single oral dose of pantoprazole
Time Frame: 1 day
Population: All patients without any major protocol violations who received 1 dose of pantoprazole on the day the PK samples were obtained, who had at least 4 blood samples, and for whom the pantoprazole terminal-phase disposition half-life could be estimated.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 17 | 18
ng/mL | 567 (534) | 1527 (1298)

2. Primary Outcome: Time to Peak Concentration (Tmax) Profile
Description: Pharmacokinetic (PK) parameters, including time to peak plasma concentration, were determined following a single oral dose of pantoprazole.
Time Frame: 1 day
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 17 | 18
hr | 1.03 [1.00 to 4.00] | 1.02 [0.50 to 4.08]

3. Primary Outcome: Disposition Half-life
Description: Pharmacokinetic (PK) parameters, including the terminal-phase disposition half-life, were determined following a single oral dose of pantoprazole. Half-life is the time required for half the quantity of absorbed drug to be metabolized or eliminated by normal biological processes.
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 17 | 18
hr | 1.78 (1.30) | 1.42 (0.78)

4. Primary Outcome: Area Under the Concentration-time Curve (AUC)
Description: Pharmacokinetic (PK) parameters, including AUC, were determined following a single oral dose of pantoprazole. AUC is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 17 | 18
ng*hr/mL | 1046 (1043) | 3602 (3269)

5. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Pharmacokinetic (PK) parameters, including apparent oral clearance, were determined following a single oral dose of pantoprazole. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr/kg
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 17 | 18
L/hr/kg | 1.54 (2.35) | 0.87 (1.36)

6. Primary Outcome: Pantoprazole Plasma Concentration After Multiple-Dose Oral Administration
Description: Plasma concentration of pantoprazole after multiple doses was measured to see if there was any accumulation of the drug.
Time Frame: 7 days
Population: All patients for whom at least 2 PK samples were obtained after 5 consecutive doses. Low dose population was 19 for both 2 and 4 hours. High dose population was 17 and 18 for 2 and 4 hours respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 19 | 18
ng/mL
  2 hours | 289 (354) | 668 (825)
  4 hours | 69 (102) | 353 (509)

7. Primary Outcome: Intragastric pH
Description: Intragastric pH is a method for evaluating gastric acidity scaled 0-9. A lower pH means more acidity. A longer duration of esophageal mucosa exposure to a gastric refluxate with a pH <4.0 correlates with more severe mucosal injury in patients with gastroesophageal reflux disease (GERD).
Time Frame: 7 days
Population: Patients who had baseline and steady-state pH-metry performed, total pH-metry recording time of at least 16 hours, and received at least 5 consecutive daily doses of pantoprazole before the steady-state pH-metry was performed.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 11 | 10
units on scale
  Baseline | 4.2 (1.4) | 3.0 (1.4)
  Steady state | 4.8 (1.3) | 4.2 (1.5)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (0.6 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.087, t-test, 2 sided; paired
Statistical Analysis 2: Comparison: High Dose Pantoprazole (1.2 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.019, t-test, 2 sided; paired

8. Primary Outcome: Median Intragastric pH
Description: as for outcome 7
Time Frame: 7 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 11 | 10
units on scale
  Baseline | 4.2 (1.7) | 2.8 (1.5)
  Steady state | 4.7 (1.7) | 4.2 (1.9)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (0.6 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.255, t-test, 2 sided; paired
Statistical Analysis 2: Comparison: High Dose Pantoprazole (1.2 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.031, t-test, 2 sided; paired

9. Primary Outcome: Percentage of Time Intragastric pH Was >4
Description: Intragastric pH is a method for evaluating gastric acidity. A lower pH means more acidity. A longer duration of esophageal mucosa exposure to a gastric refluxate with a pH <4.0 correlates with more severe mucosal injury in patients with gastroesophageal reflux disease (GERD).
Time Frame: 7 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 11 | 10
percentage of time
  Baseline | 55.5 (28.6) | 32.2 (24.1)
  Steady state | 68.5 (28.3) | 56.6 (31.1)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (0.6 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.099, t-test, 2 sided
Statistical Analysis 2: Comparison: High Dose Pantoprazole (1.2 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.016, t-test, 2 sided

10. Primary Outcome: Mean Intraesophageal pH
Description: Intraesophagel pH is a method for evaluating acidity of gastric refluxate scaled 0-9. A lower pH means more acidity. A longer duration of esophageal mucosa exposure to a gastric refluxate with a pH <4.0 correlates with more severe mucosal injury in patients with gastroesophageal reflux disease (GERD).
Time Frame: 7 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 11 | 10
units on scale
  Baseline | 5.7 (0.7) | 5.2 (0.4)
  Steady state | 5.6 (0.8) | 4.9 (0.3)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (0.6 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.347, t-test, 2 sided
Statistical Analysis 2: Comparison: High Dose Pantoprazole (1.2 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.012, t-test, 2 sided

11. Primary Outcome: Median Intraesophageal pH
Description: as for outcome 10
Time Frame: 7 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 11 | 10
units on scale
  Baseline | 5.8 (0.7) [4.7 to 7.1] | 5.3 (0.5) [4.6 to 6.0]
  Steady state | 5.6 (0.8) [4.5 to 7.3] | 4.9 (0.4) [4.5 to 5.7]
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (0.6 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.339, t-test, 2 sided
Statistical Analysis 2: Comparison: High Dose Pantoprazole (1.2 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

12. Primary Outcome: Percentage of Time That Intraesophageal pH Was <4
Description: Intraesophagel pH is a method for evaluating acidity of gastric refluxate. A lower pH means more acidity. A longer duration of esophageal mucosa exposure to a gastric refluxate with a pH <4.0 correlates with more severe mucosal injury in patients with gastroesophageal reflux disease (GERD).
Time Frame: 7 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 11 | 10
percentage of time
  Baseline | 4.6 (3.9) | 8.0 (5.6)
  Steady state | 4.6 (5.6) | 9.4 (5.8)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (0.6 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.982, t-test, 2 sided
Statistical Analysis 2: Comparison: High Dose Pantoprazole (1.2 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.534, t-test, 2 sided

13. Primary Outcome: Normalized Area of Gastric Hydrogen Ion Activity Over Time
Description: Normalized Area of Gastric Hydrogen Ion Activity Over Time is a measure of the area under the curve of the gastric hydrogen ion activity over time, which is normalized for a 24-hour period.
Time Frame: 7 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: H*mmol/L
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 11 | 10
H*mmol/L
  Baseline | 259.7 (442.7) | 921.0 (1290.1)
  Steady state | 102.3 (118.6) | 303.6 (524.9)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (0.6 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.166, t-test, 2 sided
Statistical Analysis 2: Comparison: High Dose Pantoprazole (1.2 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.119, t-test, 2 sided

14. Primary Outcome: Normalized Area of Esophageal Hydrogen Ion Activity Over Time
Description: Normalized Area of Esophageal Hydrogen Ion Activity Over Time is a measure of the area under the curve of the esophageal hydrogen ion activity over time, which is normalized for a 24-hour period.
Time Frame: 7 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: H*mmol/L
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Number analyzed (Participants) | 11 | 10
H*mmol/L
  Baseline | 2.1 (1.6) | 3.5 (2.3)
  Steady state | 1.5 (2.4) | 1.5 (0.6)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (0.6 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.387, t-test, 2 sided
Statistical Analysis 2: Comparison: High Dose Pantoprazole (1.2 mg/kg); Within group comparison between steady state and baseline; Test type: Superiority or Other; p = 0.021, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Serious Adverse Events (participants affected / at risk) | 3 | 2
Other Adverse Events (participants affected / at risk) | 13 | 17
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Gastroenteritis (Gastrointestinal disorders) | 1/33 | 1/34
Vomiting (Gastrointestinal disorders) | 1/33 | 0/34
Dehydration (Metabolism and nutrition disorders) | 1/33 | 0/34
Apnea (Respiratory, thoracic and mediastinal disorders) | 0/33 | 1/34
Stridor (Respiratory, thoracic and mediastinal disorders) | 1/33 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Low Dose Pantoprazole (0.6 mg/kg) | High Dose Pantoprazole (1.2 mg/kg)
Abdominal pain (General disorders) | 1/33 | 1/34
Fever (General disorders) | 3/33 | 4/34
Infection (General disorders) | 1/33 | 2/34
Injection site pain (General disorders) | 0/33 | 1/34
Sepsis (General disorders) | 1/33 | 0/34
Atrial septal defect (Cardiac disorders) | 1/33 | 0/34
Diarrhea (Gastrointestinal disorders) | 2/33 | 4/34
Eructation (Gastrointestinal disorders) | 1/33 | 0/34
Flatulence (Gastrointestinal disorders) | 0/33 | 2/34
Gastroenteritis (Gastrointestinal disorders) | 1/33 | 2/34
Tooth disorder (Gastrointestinal disorders) | 0/33 | 2/34
Vomiting (Gastrointestinal disorders) | 2/33 | 0/34
Creatine phosphokinase increased (Metabolism and nutrition disorders) | 1/33 | 0/34
Dehydration (Metabolism and nutrition disorders) | 1/33 | 0/34
Weight loss (Metabolism and nutrition disorders) | 0/33 | 1/34
Apnea (Respiratory, thoracic and mediastinal disorders) | 0/33 | 1/34
Cough increased (Respiratory, thoracic and mediastinal disorders) | 0/33 | 1/34
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0/33 | 1/34
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1/33 | 3/34
Contact dermatitis (Skin and subcutaneous tissue disorders) | 2/33 | 3/34
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1/33 | 0/34
Eczema (Skin and subcutaneous tissue disorders) | 0/33 | 1/34
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1/33 | 0/34
Rash (Skin and subcutaneous tissue disorders) | 1/33 | 1/34
Otitis media (Ear and labyrinth disorders) | 0/33 | 3/34
Urine abnormality (Renal and urinary disorders) | 0/33 | 1/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.